CLINICAL TRIAL: NCT05404984
Title: Effects of Core Stabilization Exercises With and Without Dry Cupping on Pain and Disability in Patients With Sacroiliac Joint Dysfunction
Brief Title: Effects of Core Stabilization Exercises With and Without Dry Cupping in Patients With Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0105
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: dry cupping; core stabilization exercise; sacroiliac joint dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry cupping with core stabilization exercises (Experimental): On 12 patients, dry cupping will be performed by using a disposable manual cupping set including a hand suction pump and plastic cups of different sizes. These cups will be placed over the points GB 30, Huantiao, BL-28 Pangguangshu, BL-54 ZHIBIAN and EM-Yaoyan. After dry cupping session core stabilization exercises will be added.
  Interventions: Other: Dry cupping with core stabilization exercises
- Core stabilization exercises (Active Comparator): 12 patients will be asked to perform core stabilization exercises where the local stabilizers of the lumbopelvic region will be targeted to ensure segmental control in different positions such as supine, crook-lying, side-lying, prone, four-point kneeling, sitting, and standing.
  Interventions: Other: Core stabilization exercises

INTERVENTIONS:
Other: Dry cupping with core stabilization exercises — 12 patients will receive dry cupping technique for 10 minutes followed by 10 repetitions of each core stabilization exercise in different positions. All the patients will receive this treatment once a week for 6 weeks.
  Arms: Dry cupping with core stabilization exercises
Other: Core stabilization exercises — A total of 12 patients will perform 10 repetitions of each core stabilization exercise in different positions. All the patients will receive this treatment once a week for 6 weeks.
  Arms: Core stabilization exercises

SUMMARY:
The aim of this study is to compare the effects of core stabilization exercises with and without dry cupping on pain and disability in patients with sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
Low back pain (LBP) is recognized by its most common symptom - pain - and is known as the primary cause of disability one of the most frequent pain-producing factors in patients with LBP is sacroiliac joint dysfunctions (SJD). The sacroiliac joint dysfunction syndrome (SIJDS) is a contentious topic that is a common cause of low back pain (LBP) and patients often seek physical therapy helps to deal with their symptoms. Dry cupping on the SIJ is a physical therapy technique that has been supported by research in numerous areas, including pain reduction and SIJ mobility promotion.

But, in previous studies, there is very less literature regarding determining effects of the dry cupping on sacroiliac joint dysfunction. Therefore there is a dire need to explore the effect of dry cupping on sacroiliac joint dysfunction. This study aims the management of pain disability and functional impairment in persons with sacroiliac joint dysfunction particularly core stabilization exercises along with dry cupping therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain for more than 3 months
* Pain on performing pain provocative tests for sacroiliac dysfunction
* Oswestry disability index above 20% but below 80%

Exclusion Criteria:

* Participants suffering from specific low back pain like PIVD with instability or any radicular symptoms, lumbar spondylosis, lumbarcanal stenosis, spondylolisthesis, sensory deficits, malignancies and tuberculosis.
* Any traumatic conditions around the pelvis and lower limbs, any infectious, tumors conditions around the pelvis.
* Pregnancy, any lower limb abnormalities, any recently underwent abdominal and low back surgery.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 6th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Modified ODI for disability | 6th week
  It is a disease-specific disability measure and is used to find the level of disability with the help of questions asking about difficulty in performing activities of daily life in 10 different sections.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. M Anbar ARA, Saleh AM, Ismail NM, El-Shazly U. CUPPING VERSUS KINESIOTAP ON MANAGEMENT OF PATIENTS WITH SACROILIAC JOINT DYSFUNCTION:"A RANDOMIZED CONTROLLED TRIAL". Delta University Scientific Journal. 2020;3(2):21-32.
- [Background] Dogan N, Sahbaz T, Diracoglu D. Effects of mobilization treatment on sacroiliac joint dysfunction syndrome. Rev Assoc Med Bras (1992). 2021 Jul;67(7):1003-1009. doi: 10.1590/1806-9282.20210436. PMID 34817514
- [Background] 7. Al-Qudah M, Khalid A-J. Impact Of Cupping Massage and Modified Spinal Decompression Therapy With Core Stabilization Exercise In Lumbar Bulging Disc Management. Psychology and Education Journal. 2021;58(3):1978-86.
- [Background] Nasb M, Qun X, Ruckmal Withanage C, Lingfeng X, Hong C. Dry Cupping, Ischemic Compression, or Their Combination for the Treatment of Trigger Points: A Pilot Randomized Trial. J Altern Complement Med. 2020 Jan;26(1):44-50. doi: 10.1089/acm.2019.0231. Epub 2019 Oct 3. PMID 31580695
- [Background] Wood S, Fryer G, Tan LLF, Cleary C. Dry cupping for musculoskeletal pain and range of motion: A systematic review and meta-analysis. J Bodyw Mov Ther. 2020 Oct;24(4):503-518. doi: 10.1016/j.jbmt.2020.06.024. Epub 2020 Jul 30. PMID 33218554
- [Background] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992
- [Background] Teut M, Ullmann A, Ortiz M, Rotter G, Binting S, Cree M, Lotz F, Roll S, Brinkhaus B. Pulsatile dry cupping in chronic low back pain - a randomized three-armed controlled clinical trial. BMC Complement Altern Med. 2018 Apr 2;18(1):115. doi: 10.1186/s12906-018-2187-8. PMID 29609566
- [Background] Kamali F, Zamanlou M, Ghanbari A, Alipour A, Bervis S. Comparison of manipulation and stabilization exercises in patients with sacroiliac joint dysfunction patients: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):177-182. doi: 10.1016/j.jbmt.2018.01.014. Epub 2018 Jan 31. PMID 30691749
- [Background] Akbarzade M, Ghaemmaghami M, Yazdanpanahi Z, Zare N, Mohagheghzadeh A, Azizi A. Comparison of the Effect of Dry Cupping Therapy and Acupressure at BL23 Point on Intensity of Postpartum Perineal Pain Based on the Short Form of McGill Pain Questionnaire. J Reprod Infertil. 2016 Jan-Mar;17(1):39-46. PMID 26962482
- [Background] Polly DW, Swofford J, Whang PG, Frank CJ, Glaser JA, Limoni RP, Cher DJ, Wine KD, Sembrano JN; INSITE Study Group. Two-Year Outcomes from a Randomized Controlled Trial of Minimally Invasive Sacroiliac Joint Fusion vs. Non-Surgical Management for Sacroiliac Joint Dysfunction. Int J Spine Surg. 2016 Aug 23;10:28. doi: 10.14444/3028. eCollection 2016. PMID 27652199
- [Derived] Noor Ul Ain; Bashir MS, Noor R, Ikram M, Iftikhar A, Najm R. Effects of core stabilisation exercises with and without dry cupping on pain and disability in patients with sacroiliac joint dysfunction. J Pak Med Assoc. 2025 Jan;75(1):61-65. doi: 10.47391/JPMA.8289. PMID 39828829